CLINICAL TRIAL: NCT07274592
Title: The Effect of Psychoeducation Program Applied to Older Adults Based on Psychosocial Development Theory on Self-critical Rumination, Self-esteem and Psychological Well-being
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Hatice Bozkaya, Nurse, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 26003
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Older Adults (65 Years and Older)
Keywords: older adults; self-esteem; rumination; psychological well-being; randomized controlled trial
MeSH Terms: conditions — Rumination Syndrome; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A standardized mini mental test will be administered to determine the inclusion criteria for non-rehabilitated elderly adults living in nursing homes. After administering pre-tests to the elderly adults, they will be assigned to the intervention and control groups using a simple randomization method. Elderly adults with a standardized mini mental test score of 25 or above on the https://www.randomizer.org/ will be assigned a number and randomized. Twenty-six individuals will be assigned to the intervention group and 26 to the control group. Randomization will be performed by the thesis advisor, and the researcher will have access to the information in the control and intervention groups prior to implementation. Support will be obtained from an independent statistician for the statistical analysis of the data in the reporting. This will prevent the risk of bias in the results.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): A standardized mini mental test will be administered at the beginning of the study to determine the inclusion criteria. Sociodemographic Information Form, Self-Critical Rumination Scale, Psychological Well-Being Scale for Older Adults, and Rosenberg Self-Esteem Scale will be applied to the control group. No intervention will be made. Measurement tools will be applied for the posttest.
- Psychoeducation Program (Experimental): A standardized mini mental test will be administered at the beginning of the study to determine the inclusion criteria. Sociodemographic Information Form, Self-Critical Rumination Scale, Psychological Well-Being Scale for Older Adults, and Rosenberg Self-Esteem Scale will be applied to pretest. The psychoeducation will be conducted once a week (on a day deemed appropriate and recommended by the nursing home) by a researcher (graduate student) with three groups. Eight sessions, each lasting 45 minutes, are planned. At the end of the sessions, post-tests of the measurement tools will be performed.
  Interventions: Behavioral: Psychoeducation Program

INTERVENTIONS:
Behavioral: Psychoeducation Program — The Psychoeducation Program, grounded in Erikson's Psychosocial Theory, is designed to help older adults cope with self-critical ruminative thoughts and improve their psychological well-being and self-esteem. Based on Erikson's eight stages of development, this program aims to help older individuals review their life journeys and understand how they experienced crises at each stage. Throughout the program, participants are encouraged to reframe their past experiences in a positive way, increase their current well-being, and strengthen their self-esteem. Older adults may face more challenges with past experiences and uncertainties about the future as they progress through life. During this process, repetitive thoughts, i.e., negative or worrisome thoughts that constantly occupy the mind, can negatively affect individuals' mental health. Psychoeducation programs are an important tool for developing coping skills for such thoughts and improving individuals' quality of life.
  Arms: Psychoeducation Program

SUMMARY:
The aim is to examine the effect of a psychoeducation program based on the Psychosocial Development Theory applied to older adults on self-critical rumination, self-esteem, and psychological well-being, as well as the relationship between these concepts. The constant and repetitive thinking of older adults about their past mistakes and failures is defined as self-critical rumination, which can have negative effects on mental health, lead to a decline in quality of life, and cause older adults to experience an unhappy process. For this study, a psychoeducation program based on Erikson's psychosocial stages of development was prepared. The program aims to differentiate rumination levels among older adults, provide suggestions on how to reduce these ruminative thoughts, and teach techniques for dealing with repetitive thoughts, thereby equipping individuals with methods to cope with ruminative thinking. It is expected that elderly individuals who acquire this coping method will experience changes in their psychological well-being and self-esteem. This study's examination of the effects of the psychoeducational program on psychological well-being provides a critical contribution to improving the quality of life of elderly individuals.

DETAILED DESCRIPTION:
This research is designed as a randomized controlled trial. The reporting of the research will be structured according to the CONSORT checklist. The Psychoeducational Program, grounded in Erikson's Psychosocial Theory, is designed to help older adults cope with self-critical ruminative thoughts and improve their psychological well-being and self-esteem. Based on Erikson's eight stages of development, this program aims to help older individuals review their life journeys and understand how they experienced crises at each stage. Throughout the program, participants are encouraged to reframe their past experiences in a positive way, increase their current well-being, and strengthen their self-esteem. Older adults may face more of their past experiences and uncertainties about the future in the later stages of their lives. During this process, repetitive thoughts, i.e., negative or worrisome thoughts that constantly occupy the mind, can negatively affect individuals' mental health. Psychoeducation programs are an important tool for developing coping skills for such thoughts and improving individuals' quality of life.

The research is planned to be conducted at Dr. İsmail Işık Retirement and Rehabilitation Center in Konya province. The sample size calculation for the study was carried out using the G*Power 3.1.9.7 program. It was calculated that a total of 48 adults, would be sufficient, with an effect size of 0.96, 95% test power, and a margin of error of 0.05. Considering the possibility of data loss in the study, the sample size was increased by 10% to include 52 older adults. The Standardized Mini Mental Test will be administered to the elderly to determine the inclusion criteria. Individuals over the age of 65, who are literate, have a Standardized Mini Mental Test score of 25 or higher, have no cognitive or perceptual problems, and volunteer to participate in the study will be included. This study also planned to use the Sociodemographic Information Form, the Self-Critical Rumination Scale, the Psychological Well-Being Scale for the Elderly, and the Rosenberg Self-Esteem Scale. The psychoeducation program consists of eight sessions. Each session will be held face-to-face once a week for the intervention group. The sessions will be conducted by a researcher (graduate student) once a week (on a day deemed appropriate and recommended by the nursing home) in three groups. Eight 45-minute sessions are planned. During their graduate studies, the researcher has acquired theoretical knowledge about psychoeducation as well as practical knowledge about its application based on the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older,
* Being literate,
* Scoring 25 or above on the Standardized Mini Mental Test,
* Having no hearing or vision problems,
* Volunteering to participate in the study

Exclusion Criteria:

* Not attending more than two psychoeducation sessions,
* Not wishing to continue the study,
* Being unable to attend due to any physical or mental health condition.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
The effect of the psychoeducation program on self-critical rumination, psychological well-being, and self-esteem | At the beginning of the study and at the end of the 8th week
  Self-Critical Rumination Scale: The Self-Critical Rumination Scale was created to determine individuals' self-critical rumination. Developed by Smart et al. (2016), the scale was adapted to Turkish by Kocalar (2019). It is a four-point Likert-type measurement tool. The scale has a 10-item, single-factor structure. There is no reverse scoring for the scale items. (Kocalar, 2019).
  Psychological Well-Being Scale in the Elderly: Developed by Gümüş Demir (2023) to measure the levels of psychological well-being in elderly individuals, the scale consists of 15 items. It is a five-point Likert-type scale. Questions 8 and 13 are reverse-coded, and the minimum score is 15 and the maximum score is 75. As the psychological well-being score increases, so does the level of well-being.
  Rosenberg Self-Esteem Scale: The scale, developed by Rosenberg (1963), was adapted into Turkish by Çuhadaroğlu (1986). The 10-item scale is rated as "very true," "true," "false," and "very false."

SECONDARY OUTCOMES:
The Effect of Psychoeducation Program Applied to Older Adults Based on Psychosocial Development Theory on Self-critical Rumination, Self-esteem and Psychological Well-being | At the beginning of the study
  Sociodemographic Information Form: This form was created by the researcher by reviewing the literature (Akgöz, 2024; Önder, 2021). There are a total of 9 questions, including age, gender, marital status, number of children, educational status, how long the patient has been staying in a nursing home, how many rooms the patient has stayed in, the reason for staying in the nursing home (own request or family request), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Adeviye AYDIN, Study Director — Necmettin Erbakan University
Locations (1):
- Dr. İsmail Işık Retirement and Rehabilitation Center, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No